CLINICAL TRIAL: NCT06979323
Title: The IMAGINE Study: A Phase 3b Open Label, Single Arm Study to Assess the Effect of Depemokimab on Airway Structure and Function in Asthma With Type 2 Inflammation Characterized by an Eosinophilic Phenotype Utilizing Quantitative High-resolution CT and Bronchoscopic Airway Sampling in a Sub Study
Brief Title: Depemokimab Asthma Imaging and Bronchoscopy Sub-Study
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 223529; 2024-519976-19 (Other: EU CT Number)
Record Dates: First submitted 2025-05-16; First posted 2025-05-18 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Asthma
Keywords: Depemokimab; Asthma; Type 2 Inflammation; Eosinophilic Phenotype; High Resolution Computed Tomography (HRCT); Bronchoscopy; IMAGINE study
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: This is a single arm study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Depemokimab (Experimental): Participants with asthma with type 2 inflammation will receive depemokimab.
  Interventions: Biological: Depemokimab

INTERVENTIONS:
Biological: Depemokimab — Depemokimab will be administered.

SUMMARY:
Asthma is a chronic condition marked by narrowed and swollen airways due to inflammation leading to recurring symptoms that can vary and worsen unpredictably. The purpose of this study is to assess how depemokimab, a monoclonal antibody, affects the structure and function of the lungs in asthmatic participants with type 2 inflammation, characterized by an eosinophilic phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Documented physician diagnosis of asthma for greater than or equal to (>=) 2 years as per the National Heart, Lung, and Blood Institute guidelines (NHLBI, 2020) or GINA guidelines along with the following: A T2 phenotype as evidenced by a blood eosinophil count of >=300 cells/microliters (mcL) at screening or a documented history of blood eosinophil count >=300 cells/mcL within 3 months prior to screening and Exhaled nitric oxide (FeNO) measure of >=25 parts per billion (ppb) recorded at screening;
* >= 2 exacerbations requiring treatment with systemic corticosteroid (SCS; intramuscular [IM], intravenous [IV], or oral), in the 12 months prior to screening, despite the use of medium to high dose Inhaled corticosteroids (ICS)
* Uncontrolled asthma indicated by Astha Control Questionnaire-5 (ACQ-5) greater than (>) 1.5 recorded at screening
* Persistent airflow obstruction as indicated by pre-bronchodilator Forced Expiration Volume in 1 second (FEV1) less than (<) 80 percentage (%) predicted (GLI 2012) and recorded at screening
* A well-documented requirement for regular treatment with medium or high dose ICS (in the 12 months prior to screening with or without maintenance oral corticosteroids [OCS])
* Current treatment with at least one additional asthma controller medication, besides ICS, for at least 3 months [for example, Long-acting Beta 2 agonists [LABA], Long-acting muscarinic antagonists [LAMA], leukotriene receptor antagonist (LTRA), or theophylline]
* Male Participants: No additional requirements for male participants
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies: is a woman of non-childbearing potential (WONCBP) or is a woman of childbearing potential (WOCBP) and using a contraceptive method that is highly effective (with a failure rate of <1% per year), with low user dependency,
* A WOCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) within 24 hours before the first dose of study intervention
* Capable of giving written informed consent,
* For the biopsy sub study participants who sign the Informed Consent for the bronchoscopy sub study, the following additional eligibility criteria will apply:

  * Participants not on maintenance OCS (oral corticosteroids) at the time of screening.
  * Participants with post bronchodilator FEV1 >= 50% predicted
  * Participants with no known increased risk for bleeding or clotting abnormalities including: No history of easy bleeding, bruising or known bleeding diathesis; No current anticoagulant and antiplatelet therapy; No acetylsalicylic acid use within 2 weeks of the planned procedure; Normal screening platelet count
  * Participants with no specific contraindication to bronchoscopy with endobronchial biopsy in the opinion of the investigator
  * No history of allergic reaction to local anesthesia or general anesthetic agent, whichever is relevant to the procedure being performed

Exclusion Criteria:

* Presence of a known pre-existing, clinically important lung condition other than asthma. This includes (but is not limited to) current infection, bronchiectasis, pulmonary fibrosis, bronchopulmonary aspergillosis, or a history of lung cancer. Participants with current diagnoses of emphysema or chronic bronchitis (Chronic obstructive pulmonary disease [COPD] other than asthma) are excluded
* Participants with other conditions that could lead to elevated eosinophils such as hyper eosinophilic syndromes including (but not limited to) Eosinophilic Granulomatosis with Polyangiitis (EGPA, formerly known as Churg-Strauss Syndrome) or eosinophilic esophagitis
* Participants who developed an exacerbation within 4 weeks before screening
* Participants with a known, pre-existing parasitic infestation within 6 months prior to screening unless treated and evidenced to have been resolved
* A known immunodeficiency (e.g. human immunodeficiency virus HIV), other than that explained by the use of corticosteroids (CSs) taken as therapy for asthma
* A current malignancy or previous history of cancer in remission for less than 12 months prior to screening
* Participants who have known, pre-existing, clinically significant cardiac, endocrine, autoimmune, metabolic, neurological, psychiatric, renal, gastrointestinal, hepatic, hematologic or any other system abnormalities that are uncontrolled with standard treatment
* Participants with current diagnosis of vasculitis
* Participants who have received mepolizumab, reslizumab, or benralizumab within 12 months prior to screening or who have a previous documented failure with anti-IL-5/5R therapy
* Participants who have received omalizumab (Xolair), dupilumab (Dupixent) or tezepelumab (Tezspire) within 12 months prior to the screening
* Participants who have received any monoclonal antibody (mAb) within 5 half-lives of the drug prior to the screening. Authorized treatments for Coronavirus disease-2019 (COVID-19) are permitted
* Participants who have received treatment with an investigational drug within the past 30 days or 5 terminal phase half-lives of the drug whichever is longer, prior to the first dose of study intervention (this also includes investigational formulations of marketed products)
* Previously participated in any clinical study with biologic treatments for asthma (for example, omalizumab, mepolizumab, dupilumab, reslizumab, benralizumab, other mAbs (including Tezepelumab) or depemokimab and received study intervention (including placebo) within 12 months prior to the first dose of study intervention
* A history (or suspected history) of alcohol misuse or substance abuse within 2 years prior to the first dose of study intervention
* Current smokers or former smokers with a smoking history >=20 pack years (number of pack years = [number of cigarettes per day/20] x number of years smoked) and vapers
* Participants with allergy/intolerance to a mAb or biologic or any of the excipients of depemokimab
* Participants who are pregnant or breastfeeding
* Participants who have known evidence of lack of adherence to controller medications and/or ability to follow physician's recommendations
* Participants who have occupational ionizing-radiation exposure exceeding 10 Millisievert (mSV) over 3 years as documented with a dosimeter; have been exposed to elevated ionizing radiation from research imaging studies, for example, Participation in a research study with a single positron emission tomography scan in the past 3 years, and Participation in a research study with 2 or more computed tomography (CT) scans in the past 3 years in the following anatomical regions: chest, abdomen, cardiac, or spine
* Presence of metal objects that may interfere with chest CT quantification including presence of a cardiac pacemaker, defibrillator, metal prosthetic heart valve, metal projectile or metal weapon fragment (bullet, shrapnel, shotgun shot) or metal shoulder prosthesis
* Evidence of clinically significant abnormality in the hematological, biochemical or urinalysis screen at screening (Visit 0), as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2028-02-11 (Estimated); Study Completion 2028-02-11 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline in Total Mucus Plug Volume Measured at Total Lung Capacity (TLC) at Week 26 | From Baseline up to Week 26
  Mean change from baseline in total mucus plug volume measured at TLC at Week 26 will be assessed.

SECONDARY OUTCOMES:
Mean Change from Baseline in Airway Wall Thickness Measured at TLC at Week 52 | From Baseline up to Week 52
  Mean change from baseline in airway wall thickness measured at TLC at Week 52 will be assessed.
Mean Change from Baseline in Airway Wall Thickness Measured at TLC at Week 26 | From Baseline up to Week 26
  Mean change from baseline in airway wall thickness measured at TLC at Week 26 will be assessed.
Mean Change from Baseline in Total Mucus Plug Volume Measured at TLC at Week 52 | From Baseline up to Week 52
  Mean change from baseline in total mucus plug volume measured at TLC at Week 52 will be assessed.
Mean Change from Baseline at Week 26 for Mucus Segment Score | From Baseline up to Week 26
  Mean change from baseline at Week 26 for mucus segment score will be assessed. The airway is divided into segments and each segment is given a score depending on the presence and severity of mucus. The segments are scored individually and then these scores are summed to give a total mucus score. (A mucus segment score between 0 - 4 indicates low levels of mucus production and a mucus segment score of 5 indicates higher levels of mucus production.)
Mean Change from Baseline at Week 52 for Mucus Segment Score | From Baseline up to Week 52
  Mean change from baseline at Week 52 for mucus segment score will be assessed. The airway is divided into segments and each segment is given a score depending on the presence and severity of mucus. The segments are scored individually and then these scores are summed to give a total mucus score. (A mucus segment score between 0 - 4 indicates low levels of mucus production and a mucus segment score of 5 indicates higher levels of mucus production.)
Mean Change from Baseline in Pre- and Post- Bronchodilator Forced Expiration Volume in 1 second (BD FEV1) at Week 26 | From Baseline up to Week 26
  Mean change from baseline in Pre- and Post- BD FEV1 at Week 26 will be assessed.
Mean Change from Baseline in Pre- and Post-BD FEV1 at Week 52 | From Baseline up to Week 52
  Mean change from baseline in Pre- and Post-BD FEV1 at Week 52 will be assessed.
Number of Participants with Adverse Events (AE) | Up to Week 65 (End of Study)
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
Number of Participants with Serious Adverse Events (SAE) | Up to Week 65 (End of Study)
  Any untoward medical occurrence resulting in death, life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, congenital anomaly/birth defect, possible drug-induced liver injury or any other situation according to medical or scientific judgment that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent serious outcomes were categorized as SAE. Number of participants who had at least one SAE or non-SAE are presented.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Plantation, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/